CLINICAL TRIAL: NCT01196169
Title: Daptomycin Use For Prophylaxis In Prosthetic Joint Surgery, A Randomized Prospective Study Comparing The Efficacy Of Daptomycin Versus Vancomycin For Peri-Operative Antibiotic Prophylaxis In MRSA Colonized Adult Patients Undergoing Primary Elective Hip, Knee or Shoulder Arthroplasty
Brief Title: Daptomycin Use for Antimicrobial Prophylaxis in Methicillin Resistant Staphylococcus Aureus (MRSA) Colonized Adult Patients Undergoing Primary Elective Hip, Knee, or Shoulder Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is closed to accrual. Enrollment of new patients stopped at the request of CUBIST Pharmaceuticals due to slow rate of enrollment.
Sponsor: Mountain Home Research & Education Corporation (Other)
Collaborators: East Tennessee State University (Other); Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0310.7f
Record Dates: First submitted 2010-06-04; First posted 2010-09-08 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Staphylococcal Infections; Methicillin-resistant Staphylococcus Aureus
Keywords: daptomycin; vancomycin; perioperative; prophylaxis; arthroplasty; prosthesis; preoperative
MeSH Terms: conditions — Staphylococcal Infections | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daptomycin (Experimental): Half of patients anticipated to be enrolled will receive daptomycin in antimicrobial prophylaxis prior to their prosthetic joint surgery.
  Interventions: Drug: Daptomycin
- Vancomycin (Active Comparator): Half of patients anticipated to be enrolled will receive vancomycin in antimicrobial prophylaxis prior to their prosthetic joint surgery.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin — One dose of Daptomycin 6 mg/Kg iv, will be infused over 30 minutes. The infusion will start no longer than one hour prior to surgical incision of primary knee or hip prosthetic joint arthroplasty.
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Vancomycin — Two doses of vancomycin 15 mg/Kg iv, with a maximum of 2 grams with each dose be infused over 60-120 minutes according to the dose. The first dose infusion will start no longer than one hour (if ≤ one gram), or no longer than two hours (if > one gram) prior to surgical incision of primary knee or hip prosthetic joint arthroplasty. A second similar dose will be given 12 hours after the first dose unless the patient has a creatinine clearance of < 50 ml/min. Patients with creatinine clearance of < 50 ml/min will only receive one dose.
  Arms: Vancomycin

SUMMARY:
This study will evaluate the safety and effectiveness of daptomycin, an antibiotic compared to another one which is vancomycin when given around the time of joint replacement surgery. Vancomycin is recommended for perioperative prophylaxis in methicillin resistant Staphylococcus aureus (MRSA) colonized patients undergoing primary total joint arthroplasty. Daptomycin has not been recommended for this indication but it is FDA approved for treatment of MRSA blood stream and skin and soft tissue infections. Data collected during this study may support the use of daptomycin for this indication and may also be used for other research purposes that have not yet been specified.

DETAILED DESCRIPTION:
This is a phase 4 randomized open label prospective pilot study comparing the use of daptomycin versus vancomycin for peri-operative antibiotic prophylaxis in patients undergoing elective primary knee, hip or shoulder arthroplasty and are at risk for infection with methicillin resistant Staphylococcus aureus. The study population will include males and non-pregnant, non-lactating females 18 years of age or older, with history of methicillin-resistant Staphylococcus aureus infection or colonization, and undergoing primary elective hip, knee or shoulder arthroplasty. The target enrollment is 100 patients, who will be randomized to daptomycin or vancomycin in two 50 patient study groups. After signing the informed consent, patients will undergo pre-enrollment nasal screening for methicillin resistant Staphylococcus aureus to identify eligible patients. Patients with positive MRSA nasal screen will proceed with enrollment and get randomized into one of the two study groups. In one group, patients will receive one dose of daptomycin 6 mg/kg to be infused over 30 minutes. In this group, the infusion should be started and completed within 60 minutes of surgical incision. In the second group, patients will receive one dose of vancomycin 15 mg/kg to be infused over 1-2 hours of surgical incision according to the dose to avoid red man syndrome. In this group, the infusion should be started and completed within 120 minutes of surgical incision. After surgery, a second similar dose of vancomycin will be given 12 hours after the first dose to patients with creatinine clearance (CLcr.) of ≥50 ml/min. All patients in both groups will be asked to shower with chlorhexidine skin cleanser (HIBICLENS®) once daily from the neck down for 7days before surgery and apply Mupirocin ointment 2% to their nostrils twice daily for 5 days before surgery.

The patients will be evaluated on the day of surgery, at 2-3 days postoperatively, on discharge, at one month and three months follow up visits. During these study evaluations, patients will be assessed clinically for signs and symptoms of wound, and prosthetic joint infection (including pain, tenderness, swelling, erythema, poor wound healing and wound drainage) prior to hospital discharge, and at one, and three months follow up visits. Blood work including complete blood counts, erythrocytic sedimentation rate, c-reactive protein, and cultures will be ordered if clinical findings suggest infection. Bacterial isolates causing infections will be tested locally for antibiotic susceptibilities including daptomycin and vancomycin and saved for further testing if needed. Adverse effects and tolerability will be documented with the use of both drugs in the two patient groups. Data will be collected and analyzed with appropriate testing. The primary endpoint will be the success in prevention of postoperative SSI and prosthetic joint infection at one month postoperative follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed, and dated informed consent as defined by the Institutional Review Board.
* Male and female patients older than 18 years of age undergoing primary elective hip, knee or shoulder arthroplasty.
* Documented nasal carriage of MRSA.
* If a female of childbearing potential the patient should agree to practice a reliable contraceptive method (e.g. birth control pills, condoms, or intrauterine device [IUD]) during treatment and for one month after receiving the study medication.

Exclusion Criteria:

* Concurrent urinary tract infection or colonization unless treated with evidence of microbiologic cure.
* Evidence of active infection elsewhere other than urinary tract, unless treated with evidence of microbiologic cure documented by the infectious diseases service.
* Patients undergoing elective secondary arthroplasty.
* Concurrent open wounds
* Pregnant and nursing women (if patient is still of childbearing potential, a negative serum pregnancy test will be confirmed).
* History of allergy or contraindication to study drugs.
* Weight >150 kg or <50kg
* Patients with creatinine clearance (CLcr) < 30ml/min (calculated using the Cockcroft-Gault equation using ideal body weight)
* Severe neutropenia (absolute neutrophil count <0.500x103 /µl).
* Patients considered unlikely to comply with study procedures or to return for the scheduled post treatment evaluation.
* Ongoing antibiotic therapy for active infection that is anticipated to continue until the day of surgery.
* Any other condition that in the opinion of the investigator, would confound or interfere with evaluation of safety or efficacy of the investigational medication, or prevent compliance with the study protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Daptomycin efficacy in prevention of postoperative surgical site infection (SSI) | 24 months
  Efficacy of daptomycin in preventing postoperative SSI will be determined for each enrolled subject on one month postoperative visit. Overall efficacy of daptomycin among the patient group who receive it will be compared to overall efficacy of vancomycin among the second patient group who receive vancomycin upon anticipated complete enrollment study at 24 months.

SECONDARY OUTCOMES:
Efficacy of daptomycin in preventing postoperative early prosthetic joint infection | 30 months
  Efficacy of daptomycin in preventing postoperative early prosthetic joint infection will be determined for each enrolled subject on three months postoperative visit. Overall efficacy of daptomycin among the patient group who receive it will be compared to overall efficacy of vancomycin among the second patient group who receive vancomycin upon anticipated completion of the study at 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Wael E Shams, M.D., Principal Investigator — James H Quillen VA Medical Center and East Tennessee State University
Locations (2):
- United States (2):
  - Johnson City Medical Center, Johnson City, Tennessee
  - James H Quillen VA Medical Center, Mountain Home, Tennessee

REFERENCES:
- [Background] Bratzler DW, Houck PM; Surgical Infection Prevention Guidelines Writers Workgroup; American Academy of Orthopaedic Surgeons; American Association of Critical Care Nurses; American Association of Nurse Anesthetists; American College of Surgeons; American College of Osteopathic Surgeons; American Geriatrics Society; American Society of Anesthesiologists; American Society of Colon and Rectal Surgeons; American Society of Health-System Pharmacists; American Society of PeriAnesthesia Nurses; Ascension Health; Association of periOperative Registered Nurses; Association for Professionals in Infection Control and Epidemiology; Infectious Diseases Society of America; Medical Letter; Premier; Society for Healthcare Epidemiology of America; Society of Thoracic Surgeons; Surgical Infection Society. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Clin Infect Dis. 2004 Jun 15;38(12):1706-15. doi: 10.1086/421095. Epub 2004 May 26. PMID 15227616
- [Background] Zimmerli W, Trampuz A, Ochsner PE. Prosthetic-joint infections. N Engl J Med. 2004 Oct 14;351(16):1645-54. doi: 10.1056/NEJMra040181. No abstract available. PMID 15483283
- [Background] Price CS, Williams A, Philips G, Dayton M, Smith W, Morgan S. Staphylococcus aureus nasal colonization in preoperative orthopaedic outpatients. Clin Orthop Relat Res. 2008 Nov;466(11):2842-7. doi: 10.1007/s11999-008-0337-x. Epub 2008 Jun 19. PMID 18563506
- [Background] Lamp KC, Friedrich LV, Mendez-Vigo L, Russo R. Clinical experience with daptomycin for the treatment of patients with osteomyelitis. Am J Med. 2007 Oct;120(10 Suppl 1):S13-20. doi: 10.1016/j.amjmed.2007.07.010. PMID 17904946
- [Background] Marculescu CE, Osmon DR. Antibiotic prophylaxis in orthopedic prosthetic surgery. Infect Dis Clin North Am. 2005 Dec;19(4):931-46. doi: 10.1016/j.idc.2005.07.002. PMID 16297740